CLINICAL TRIAL: NCT02628054
Title: Investigating the Effects of Typhoid Vaccine on Sleep in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MSD-IDREC-C3-2014-011
Record Dates: First submitted 2015-11-19; First posted 2015-12-11 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Typhoid Vaccine on Sleep
Keywords: PSG; Typhoid Vaccine; Depression; Inflammation
MeSH Terms: conditions — Depression; Inflammation | interventions — Typhoid-Paratyphoid Vaccines; Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Typhoid Vaccine (Active Comparator): Typhoid vaccination in single 0.5mL injections into the non-dominant deltoid muscle in the arm
  Interventions: Biological: Typhoid Vaccine
- Placebo (Placebo Comparator): A single 0.5mL injection of 0.9% sodium chloride saline solution into the non-dominant deltoid muscle in the arm
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Typhoid Vaccine — Typhoid Vaccine injection given 7 days apart
  Other Names: Typhim Vi®
  Arms: Typhoid Vaccine
Biological: Placebo — Saline injection given 7 days apart
  Other Names: 0.9% sodium chloride saline solution
  Arms: Placebo

SUMMARY:
Research studies have found a relationship between the immune system (how the body reacts to an infection) and the development of depression. As it is still unclear how they might be linked the investigators will use a typhoid vaccination to activate the body's immune system and will measure the response by looking at changes in sleep patterns.

DETAILED DESCRIPTION:
Elevated levels of pro-inflammatory cytokines are implicated in the pathogenesis of major depression. Both clinical and animal studies have shown that pro-inflammatory cytokines can induce a behavioural repertoire of symptoms collectively referred to as 'sickness behaviours,' which include cognitive and mood symptoms, such as depression, anxiety, memory impairment, fatigue, anhedonia and sleep disturbance.

Raised circulating pro-inflammatory cytokines exhibited during chronic medical illness, such as rheumatoid arthritis, are frequently associated with higher rates of co-morbid depression compared to the general population. Medically healthy individuals with major depression have also been shown to have raised pro-inflammatory cytokine levels. Moreover, administration of interferon-α (IFN-α), a recombinant form of inflammatory cytokine that is commonly used as a therapy for hepatitis C virus (HCV) and certain cancers, is well documented to precipitate depression and cognitive impairment in 30-50% of patients. In a previous study in this Department the investigators showed, using magnetic resonance spectroscopy (MRS), that IFN- α increased markers of glutamate activity. This is of particular interest because of the postulated role of glutamate in mood regulation and cognition.

Converging evidence of the link between inflammation and depression has therefore led to the hypothesis that chronic low-grade inflammation could lead to more persistent alterations in neuropsychological function that might be instrumental in the pathogenesis of major depression. However, the mechanisms for this potential modulation of mood and cognitive function remain unclear.

In order to examine the relationship between inflammation and depression, experimental models of inflammation have been developed that involve exogenous administration of cytokines or cytokine-inducers, for example salmonella typhi (typhoid) vaccination. This study will utilise typhoid vaccination as a model of acute inflammatory challenge in healthy volunteers, which has previously been shown to stimulate a mild, non-sickness inducing inflammatory response that significantly increases levels of the pro-inflammatory cytokine, interleukin (IL)-6, in a safe manner without increasing symptoms of illness, body temperature and blood pressure. This model has been shown to elicit a transient depression-like syndrome in healthy volunteers, including a range of behavioural changes such as cognitive dysfunction, fatigue and modulation of subjective ratings of mood. The investigators believe this will serve as a good model to investigate effects of immune activation on sleep.

Sleep electroencephalogram (EEG) recordings will explore the effects of immune activation on sleep, as sleep changes are observed in clinical depression. Healthy volunteers will be recruited for this study, so that the investigators can investigate the effects of inflammatory challenge in participants that do not currently have an inflammatory condition.

The present exploratory study therefore aims to enhance the investigators understanding of the intriguing link between inflammation and emotional dysfunction by examining the effects of inflammatory challenge using typhoid vaccine on sleep using a detailed psychiatric assessment and sleep EEG recordings.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Healthy adults, Male or Female, aged 18 to 40 years.
* Not currently taking any medications (except the contraceptive pill).
* Good sleeper determined by self-report and sleep screening interview

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Any current or previous Axis 1 psychiatric disorder on DSM-5
* Diagnosis of current sleep disorder
* Any significant current medical condition likely to interfere with the conduct of the study or analysis of data
* Typhoid vaccination within the last 3 years
* Any vaccination within the last 6 months
* History of allergies to drugs or vaccines or any component of the typhoid vaccine
* Congenital or acquired immune deficiency (including participants receiving immunosuppressive or antimitotic drugs)
* Bleeding disorder, e.g. haemophilia or thrombocytopenia
* Current or recent physical illness or infection within previous 2 weeks
* Steroidal or non-steroidal anti-inflammatory medication within preceding 2 weeks, including aspirin and ibuprofen
* Current substance misuse
* Child bearing age and not using reliable form of contraception
* Has taken part in a psychological or medical experiment involving taking any kinds of drugs within the last 6 weeks
* Pregnant or breast feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Acute (night 1) differences in sleep architecture, measured using polysomnography, following afternoon administration of the typhoid vaccine compared to placebo (saline) injection | 19 hours

SECONDARY OUTCOMES:
Changes in Interleukin-6 (IL-6) levels following typhoid vaccine compared to placebo (saline) injection | 2 hours
  Blood sample taken 2 hours post injection
Change in PANAS subjective mood rating scores, following afternoon administration of the typhoid vaccine compared to placebo (saline) injection | 1 hour, 2 hours, 3 hours, 4 hours
Change in VAS Bond and Lader subjective mood rating scores, following afternoon administration of the typhoid vaccine compared to placebo (saline) injection | 1 hour, 2 hours, 3 hours, 4 hours
Change in adverse effects scores, following afternoon administration of the typhoid vaccine compared to placebo (saline) injection | 1 hour, 2 hours, 3 hours, 4 hours and 19 hours
Change in LSEQ subjective rating scores, following afternoon administration of the typhoid vaccine compared to placebo (saline) injection | 19 hours
Randomisation guess, following afternoon administration of the typhoid vaccine compared to placebo (saline) injection | 19 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ann L Sharpley, BSc, PhD, Principal Investigator — Psychopharmacology Research Unit

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anisman H. Cascading effects of stressors and inflammatory immune system activation: implications for major depressive disorder. J Psychiatry Neurosci. 2009 Jan;34(1):4-20. PMID 19125209
- [Background] Brydon L, Harrison NA, Walker C, Steptoe A, Critchley HD. Peripheral inflammation is associated with altered substantia nigra activity and psychomotor slowing in humans. Biol Psychiatry. 2008 Jun 1;63(11):1022-9. doi: 10.1016/j.biopsych.2007.12.007. Epub 2008 Feb 1. PMID 18242584
- [Background] Brydon L, Walker C, Wawrzyniak A, Whitehead D, Okamura H, Yajima J, Tsuda A, Steptoe A. Synergistic effects of psychological and immune stressors on inflammatory cytokine and sickness responses in humans. Brain Behav Immun. 2009 Feb;23(2):217-24. doi: 10.1016/j.bbi.2008.09.007. Epub 2008 Sep 20. PMID 18835437
- [Background] Dantzer R, O'Connor JC, Freund GG, Johnson RW, Kelley KW. From inflammation to sickness and depression: when the immune system subjugates the brain. Nat Rev Neurosci. 2008 Jan;9(1):46-56. doi: 10.1038/nrn2297. PMID 18073775
- [Background] Felger JC, Lotrich FE. Inflammatory cytokines in depression: neurobiological mechanisms and therapeutic implications. Neuroscience. 2013 Aug 29;246:199-229. doi: 10.1016/j.neuroscience.2013.04.060. Epub 2013 May 3. PMID 23644052
- [Background] Harrison NA, Brydon L, Walker C, Gray MA, Steptoe A, Critchley HD. Inflammation causes mood changes through alterations in subgenual cingulate activity and mesolimbic connectivity. Biol Psychiatry. 2009 Sep 1;66(5):407-14. doi: 10.1016/j.biopsych.2009.03.015. Epub 2009 May 7. PMID 19423079
- [Background] Harrison NA, Brydon L, Walker C, Gray MA, Steptoe A, Dolan RJ, Critchley HD. Neural origins of human sickness in interoceptive responses to inflammation. Biol Psychiatry. 2009 Sep 1;66(5):415-22. doi: 10.1016/j.biopsych.2009.03.007. Epub 2009 May 1. PMID 19409533
- [Background] Miller AH, Maletic V, Raison CL. Inflammation and its discontents: the role of cytokines in the pathophysiology of major depression. Biol Psychiatry. 2009 May 1;65(9):732-41. doi: 10.1016/j.biopsych.2008.11.029. Epub 2009 Jan 15. PMID 19150053
- [Background] Motivala SJ, Sarfatti A, Olmos L, Irwin MR. Inflammatory markers and sleep disturbance in major depression. Psychosom Med. 2005 Mar-Apr;67(2):187-94. doi: 10.1097/01.psy.0000149259.72488.09. PMID 15784782
- [Background] Raison CL, Borisov AS, Broadwell SD, Capuron L, Woolwine BJ, Jacobson IM, Nemeroff CB, Miller AH. Depression during pegylated interferon-alpha plus ribavirin therapy: prevalence and prediction. J Clin Psychiatry. 2005 Jan;66(1):41-8. doi: 10.4088/jcp.v66n0106. PMID 15669887
- [Background] Raison CL, Capuron L, Miller AH. Cytokines sing the blues: inflammation and the pathogenesis of depression. Trends Immunol. 2006 Jan;27(1):24-31. doi: 10.1016/j.it.2005.11.006. Epub 2005 Nov 28. PMID 16316783
- [Background] Wright CE, Strike PC, Brydon L, Steptoe A. Acute inflammation and negative mood: mediation by cytokine activation. Brain Behav Immun. 2005 Jul;19(4):345-50. doi: 10.1016/j.bbi.2004.10.003. Epub 2004 Dec 8. PMID 15944074
- [Derived] Sharpley AL, Cooper CM, Williams C, Godlewska BR, Cowen PJ. Effects of typhoid vaccine on inflammation and sleep in healthy participants: a double-blind, placebo-controlled, crossover study. Psychopharmacology (Berl). 2016 Sep;233(18):3429-35. doi: 10.1007/s00213-016-4381-z. Epub 2016 Aug 9. PMID 27503474